CLINICAL TRIAL: NCT04079127
Title: A Multi-centre, Non-comparative, Retrospective Post-market Surveillance Study to Obtain Clinical Outcomes Data on the Zimmer Avenir Müller Hip Stem
Brief Title: Avenir Müller Hip Stem Post Market Surveillance Study
Status: Completed | Type: Observational
Sponsor: Zimmer Biomet (Industry)
Responsible Party: Sponsor
Other Study IDs: 09H08
Record Dates: First submitted 2019-09-02; First posted 2019-09-06 (Actual); Results first posted 2020-06-23 (Actual); Last update posted 2021-05-14 (Actual); Status verified 2021-04

CONDITIONS: Osteoarthritis, Hip; Rheumatoid Arthritis; Fracture of Hip; Dislocated Hip; Osteonecrosis; Post-traumatic; Arthrosis; Subluxation Hip
MeSH Terms: conditions — Osteoarthritis, Hip; Arthritis, Rheumatoid; Hip Fractures; Hip Dislocation; Osteonecrosis; Osteoarthritis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: FDA-regulated Drug: No

GROUPS / COHORTS (1):
- Patients suffering from severe hip pain and disability: Patients in need of a total hip arthroplasty.
  Interventions: Device: Patients who met the inclusion/exclusion criteria to receive the Avenir Müller stem.

INTERVENTIONS:
Device: Patients who met the inclusion/exclusion criteria to receive the Avenir Müller stem. — Consecutive cohort of patients enrolled at every site who received the Avenir Müller stem.

SUMMARY:
This study is a Post Market Clinical Follow up study to fulfil the post market surveillance obligations according to Medical Device Directive and European Medical Device Vigilance System (MEDDEV) 2.12-2. The data collected from this study will serve the purpose of confirming safety and performance of the Avenir Müller Hip Stem.

DETAILED DESCRIPTION:
The objective of this post market surveillance study is to obtain outcome data on the Avenir Müller Hip Stem by analysis of standard scoring systems, radiographs and adverse event records, and thus to assess the long-term performance and safety of this implant.

This is a multi-centre, retrospective post-market surveillance study involving orthopaedic surgeons skilled in hip surgery. Each case enrolled has received the Avenir Müller Hip Stem for a primary hip arthroplasty. The Avenir Müller Hip Stem is CE marked (European Conformity) and commercially available.

ELIGIBILITY:
Inclusion Criteria:

* Patients able to participate in a follow-up program based upon physical examination and medical history.
* Patients or patient's legal representatives who have given written consent to take part in the study by signing the 'Patient Consent Form'.
* 18 years minimum.
* Male and female.
* Baseline data exist (pre-, peri- and immediate postoperative)

Exclusion Criteria:

* Patients who are unwilling or unable to comply with the follow-up program.
* Known pregnancy.
* Patients who are skeletally immature.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients suffering from severe hip pain and disability requiring a total hip arthroplasty.
Sampling Method: Probability Sample
Enrollment: 150 (Actual)
Dates: Start 2010-01-09 (Actual); Primary Completion 2019-06-29 (Actual); Study Completion 2019-08-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Paola Vivoda, Study Director — Zimmer Biomet

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Erivan R, Villatte G, Brientini JM, Kreider D, Descamps S, Boisgard S. 7-year results of primary total hip arthroplasty with the uncemented Avenir stem. Hip Int. 2019 Jul;29(4):418-423. doi: 10.1177/1120700018810211. Epub 2018 Nov 11. PMID 30415580

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Patients Suffering From Severe Hip Pain and Disability
Started | 150 (hips (in 141 patients))
Completed | 89 (89 hips have completed the study, and all 10 year data of 81 were available for analysis.)
Not Completed | 61

BASELINE CHARACTERISTICS:
Groups:
- Patients Suffering From Severe Hip Pain and Disability: Patients in need of a total hip arthroplasty.
  Consecutive cohort of patients enrolled at every site who received the Avenir Müller stem and who met the study inclusion/exclusion criteria .
Arm/Group | Patients Suffering From Severe Hip Pain and Disability
Number analyzed (Participants) | 150
Age, Continuous [Mean (Standard Deviation); unit: years] | 60.5 (10.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 76
  Male | 74
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Body Mass Index (BMI) kg/m2 [Mean (Standard Deviation); unit: kg/m^2] | 27.3 (4.0)
Height (cm) [Mean (Standard Deviation); unit: cm] | 168.6 (8.8)
Weight (kg) [Mean (Standard Deviation); unit: kg] | 78.1 (14.2)

OUTCOME MEASURES:

1. Primary Outcome: Evaluation of Pain and Functional Performance Determined by the Harris Hip Score
Description: The Harris Hip Score is a questionnaire filled by the surgeon with the patient who received a hip implant. The domains covered are pain, function, absence of deformity, and range of motion. The pain domain measures pain severity and its effect on activities and need for pain medication.
  The function domain consists of daily activities (stair use, using public transportation, sitting, and managing shoes and socks) and gait (limp, support needed, and walking distance). Deformity takes into account hip flexion, adduction, internal rotation, and extremity length discrepancy. Range of motion measures hip flexion, abduction, external and internal rotation, and adduction.
  There are 10 items. The score has a maximum of 100 points (best possible outcome) covering pain (1 item, 0-44 points), function (7 items, 0-47 points), absence of deformity (1 item, 4 points), and range of motion (2 items, 5 points).
Time Frame: 10 years
Population: The HHS values are within the interval 0-100 points and the higher the score is, the better the outcome is for the individuals. The results are interpreted with the following ratings: <70 points = poor result; 70-79 points = fair, 80-89 points = good, and 90-100 points = excellent.
  Number Of Unilateral Patients: 68; Number Of Bilateral Patients:7. Here, the data at 10 year post surgery of 75 patients (82 hips) were available for analysis.
Measure: Mean (Standard Deviation); unit: score on a scale
Units Other Than Participants: Implants
Arm/Group | Patients Suffering From Severe Hip Pain and Disability
Number analyzed (Participants) | 75
Number analyzed (Implants) | 82
score on a scale | 90.9 (11.7)

2. Secondary Outcome: Confirmation of Safety Based on Complications
Description: Number of patients with adverse events related to the implant will be reported. Adverse events include: dislocations of the hip, revisions and removals of the implant components.
  Here, the entire cohort of patients (and hips) enrolled in the study were considered and are reported as the complications occured from the early stages of the study, and up to 10 year post surgery, and could occur to any patients.
Time Frame: up to 10 years
Population: Revisions due to any component (Avenir Muller Hip Stem, Acetabular Insert , Acetabular Cup...) complication.
Measure: Number; unit: Patients
Units Other Than Participants: Implants
Arm/Group | Patients Suffering From Severe Hip Pain and Disability
Number analyzed (Participants) | 141
Number analyzed (Implants) | 150
Patients | 10

3. Secondary Outcome: Survivorship of the Implant
Description: Implant survival based on removal or intended removal of the device and determined using the Kaplan-Meier method.
  Here, the entire cohort of patients (and hips) enrolled in the study were considered and are reported as the revisions could happen from the early stages of the study, and up to 10 year post surgery, and could occur to any patients. Even if a patient did not come back for a visit, the information if the implant was still in place was provided and taken into account for the survival analysis (gives higher numbers than for the clinical evaluation).
Time Frame: 10 years
Population: Kaplan-Meier survival rate at 10 years post-surgery,with Avenir Muller Hip Stem revision for any reason as endpoint.
  Number of Unilateral Patients: 88; Number of Bilateral Patients: 4. Data of 88 patients,96 hips were received up to 10 years post surgery for the survival. Indeed, if a patient did not come back for a visit, the information if the implant was still in place was provided (gives higher numbers than for the clinical evaluation).
Measure: Number; unit: percentage implant survival
Units Other Than Participants: Implants
Arm/Group | Patients Suffering From Severe Hip Pain and Disability
Number analyzed (Participants) | 92
Number analyzed (Implants) | 96
percentage implant survival | 98.54

ADVERSE EVENTS:
Time Frame: The adverse events were collected preoperatively, intraoperatively and postoperatively (at 3-4 years, 5 years, 7 years and 10 years postoperative).
Description: All the 141 patients were considered in the Adverse Events report section as any hip could have an Adverse Event at any time of the study.
Arm/Group | Patients Suffering From Severe Hip Pain and Disability
All-Cause Mortality (participants affected / at risk) | 3/141
Serious Adverse Events (participants affected / at risk) | 17/141
Other Adverse Events (participants affected / at risk) | 14/141
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Patients Suffering From Severe Hip Pain and Disability (N=141)
Fracture of Femoral Shaft (Surgical and medical procedures) | 1 — Treated by revision of the Avenir Muller Stem
Bascule Implant cotyl (Surgical and medical procedures) | 1 — Treated by revision
Post traumatic Pain on acetabular (Social circumstances) | 1
Cup pain after Trauma (Social circumstances) | 1 — Treated by revision of the Cup Head
Deep Infection (>6 Weeks (Infections and infestations) | 1 — Treated by the revision of the whole prosthesis
Cardiac Arrhythmia (Cardiac disorders) | 1 — Treated by a pacemaker
Urinary Retention (Renal and urinary disorders) | 1 — Treated with a catheter
Bascule Insert acetabular (Surgical and medical procedures) | 1 — Treated by revision of the cup head
Pulmonary Embolism (Vascular disorders) | 1
Myelofibrosis (Blood and lymphatic system disorders) | 1
Reaction Due To Metal Bearing (Immune system disorders) | 1
Metallosis (Product Issues) | 1
Calcar crack (Surgical and medical procedures) | 1
Deep Infection (>6 Weeks) (Infections and infestations) | 1 — Treated by rifadin and batrim
Scar Inflammation (Blood and lymphatic system disorders) | 1 — Treated by Amoxiciline
Death (General disorders) | 1 — Cause of Death unknown.
Stroke (Blood and lymphatic system disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Patients Suffering From Severe Hip Pain and Disability (N=141)
Polymyalgia rheumatica (Congenital, familial and genetic disorders) | 1 — Treated by medical corticosteroid.
Kidney stone (Renal and urinary disorders) | 1 — Treated by Lithotripsy
Anaemia (Blood and lymphatic system disorders) | 1 — Treated by Medication
Stroke (Blood and lymphatic system disorders) | 1 — Treated by Catheter
Cardiac Arrhythmia (Cardiac disorders) | 1 — Treated by Electrical Radioscopic Treatment
Urinary Tract Infection (Infections and infestations) | 1 — Treated by Antibiotics.
Respiratory Infection (Infections and infestations) | 1 — Treated by Antibiotics
Stroke (Blood and lymphatic system disorders) | 1 — Treated by operation
Pulmonary Embolism (Vascular disorders) | 1
Dislocation (Surgical and medical procedures) | 1 — Treated by reduction with general anaesthesia
Hodgkin's disease (Blood and lymphatic system disorders) | 1 — Treated by hospitalizations and chemotherapy
Nephrectomy L and Partiel R (Renal and urinary disorders) | 1 — Treated by surgery and hospitalization.
Instability (General disorders) | 1 — Kept under surveillance
Subluxation (Surgical and medical procedures) | 1 — Treated by hospitalisation traction Nonsteroidal anti-inflammatory drugs (NSAIDs)
Ankylosing Spondylartis (Musculoskeletal and connective tissue disorders) | 1
Dislocation (Surgical and medical procedures) | 1 — Treated by reduction traction

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2009-10-06): https://cdn.clinicaltrials.gov/large-docs/27/NCT04079127/Prot_SAP_001.pdf